CLINICAL TRIAL: NCT06926543
Title: Phase III Randomized Controlled Trial of Sequential Chemotherapy and Radiotherapy Versus Concurrent Chemoradiotherapy in Adjuvant Treatment of Breast Cancer (CONCERT)
Brief Title: Postoperative Radiotherapy in Breast Cancer- Concurrent or Sequential With Chemotherapy
Acronym: CONCERT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Tabassum Wadasadawala (Other)
Responsible Party: Sponsor-Investigator, Dr. Tabassum Wadasadawala, Professor and Radiation oncologist, Tata Memorial Centre
Organization: Tata Memorial Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4131; CTRI/2023/06/054280 (Registry Identifier: Clinical Trials Registry - India (ICMR-NIMS))
Record Dates: First submitted 2025-02-14; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Invasive Breast Cancer; Stage III Breast Cancer; Stage IIB Breast Cancer
Keywords: Invasive breast cancer; Chemoradiation; Sequential; Concurrent; adjuvant therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Standard Arm (Active Comparator): Participants randomized to arm A arm will receive sequential chemotherapy and radiotherapy
  Interventions: Drug: Chemoradiation
- Arm B: Experimental arm (Experimental): Participants randomized to arm B will receive concurrent chemotherapy and radiotherapy
  Interventions: Drug: Chemoradiation

INTERVENTIONS:
Drug: Chemoradiation — This intervention will consist of getting chemotherapy followed by radiotherapy, i.e, in a sequential manner
  Arms: Arm A: Standard Arm
Drug: Chemoradiation — This intervention will consist of getting chemotherapy and radiotherapy at the same time, i.e, in a concurrent manner.
  Arms: Arm B: Experimental arm

SUMMARY:
This clinical research aims to determine if concurrent chemotherapy and radiation therapy is more effective than sequential chemotherapy and radiation therapy for patients with stage IIB-III breast cancer. It seeks to answer the following key questions:

1. When compared to sequential treatment, does concurrent chemoradiotherapy increase disease-free survival?
2. What effects does concurrent treatment have on post-operative look, quality of life, and side effects including arm swelling (lymphoedema)?
3. What are each treatment approach's financial costs?

Researchers will compare the following to groups:

Arm A: Participants in the sequential treatment group will first undergo chemotherapy and then radiation.

and Arm B: Participants in the concurrent treatment group will undergo radiation therapy while undergoing chemotherapy.

Participants are going to:

1. Get the usual chemotherapy (taxanes and/or anthracyclines).
2. Receive radiation therapy for three to four weeks.
3. Have follow-up visits every 6months for 5years to check for cancer recurrence, side effects, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed invasive breast cancer
2. Stage IIB-III invasive breast cancer (AJCC 8th edition)
3. Patients planned for adjuvant chemotherapy and adjuvant radiotherapy
4. Patients fit to receive adjuvant chemotherapy and radiotherapy
5. Age > 18 years

Exclusion Criteria:

1. Hypersensitivity to taxanes
2. Patients receiving entire chemotherapy prior to surgery (neoadjuvant setting)
3. Unable or unwilling for regular follow up
4. Bilateral tumour needed RT to both sides
5. Patients planned for RT to oligometastatic sites
6. Unfavourable anatomical factors potentially leading to higher radiotherapy dose to heart and/or lungs (Exceeding the protocol specific mandatory dose constraints).
7. Pregnant patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 858 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2031-05 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Study the 3-year Disease Free Survival. | From enrollment to 3 years after treatment at six months intervals.

SECONDARY OUTCOMES:
Impact of concurrent regimen on patient's Quality of life using the EORTC QLQ 30 and BR 23 and EQ5D5L questionnaire. | From enrollment at pre-raditherapy, post-radiotherapy completion and on follow up at 12-monthly interval up to 3 years.
Subjective and objective assessment of cosmesis in breast-conserving surgery patients, utilizing the Harvard scale and the BCCT core photographic evaluation, respectively. | From enrollment at pre-raditherapy, post-radiotherapy completion and on follow up at 12-monthly interval up to 3 years.
  All patients who undergo breast conservation surgery will be eligible for this sub-study in which we intend to collect frontal breast photographs for objective assessment of breast cosmesis.
The difference in direct and indirect cost of treatment in the two arms will be assessed using the FACT-COST. | From enrollment at start of adjuvant chemotherapy, pre-radiotherapy and at post radiotherapy treatment.
  As patients in the intervention arm will complete their treatment at least 6-8 weeks before the patients in the standard arm, it will have huge impact on the expenditure that the patient bears for staying, food as well as transport to the hospital. Hence, we would like to collect data pertaining to patient's daily expenditure during their adjuvant treatment.
To assess the rate of lymphedema in the two arms of the trial using subjective and objective methods | From enrollment at pre-radiotherapy, post-radiotherapy completion and annually thereafter till 3 years
  As the breast cancer treatment increases the risk of swelling in the upper limb, we would like to assess for the same. This will help us to diagnose lymphedema at an early stage and will be able to treat it more effectively.
Overall survival (OS)outcome assessment in the two arms. | From enrollment to 5 years after treatment at 6 months intervals
Breast Cancer Specific Survival (BCSS) will be assessed with regular follow-ups. | From enrollment to 5 years after treatment at 6 months intervals

CONTACTS AND LOCATIONS:
Locations (5):
- India (5):
  - Homi Bhabha Cancer Hospital & Research Centre, Vishkhapatnam, Andhra Pradesh
  - Tata Memorial Centre, Mumbai, Maharasthra
  - Homi Bhabha Cancer Hospital and Research Centre, New Chandigarh, Punjab
  - Homi Bhabha Cancer Hospital, Sangrur, Sangrur, Punjab
  - Mahamana Pandit Madan Mohan Malviya Cancer Centre, Varanasi, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wadasadawala T, Anup A, Carlton J, Sarin R, Gupta S, Parmar V, Pathak R, Ghosh J, Bajpai J, Gulia S, Krishnamurthy R. CONcurrent ChEmotherapy and RadioTherapy in adjuvant treatment of breast cancer (CONCERT): a phase 2 study. Ecancermedicalscience. 2023 Feb 23;17:1510. doi: 10.3332/ecancer.2023.1510. eCollection 2023. PMID 37113709
- See also: A Pilot Study of CONcurrent ChEmotherapy and RadioTherapy in Adjuvant Treatment of Breast Cancer (CONCERT) — https://ecancer.org/en/journal/article/1510-concurrent-chemotherapy-and-radiotherapy-in-adjuvant-treatment-of-breast-cancer-concert-a-phase-2-study